CLINICAL TRIAL: NCT06208254
Title: Prevalence and Risk Indicators of Peri-implant Diseases in China: A Multicenter Cross-sectional Study
Brief Title: Prevalence and Risk Indicators of Peri-implant Diseases in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Collaborators: Dalian Medical University (Other); Nanchang University (Other); Ningxia Medical University (Other); Shanxi Medical University (Other); Hospital of Stomatology, Wuhan University (Other); Hospital of Stomatology, Sun Yat-Sen University (Other); Zunyi Medical College (Other); Hong Kong Brånemark Osseointegration Center (Other)
Responsible Party: Sponsor
Other Study IDs: SDC-23-3
Record Dates: First submitted 2024-01-03; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients having at least one rough surface titanium implant in function for more than 5 years.

SUMMARY:
The goal of this multicenter cross-sectional study is to investigate the prevalence of peri-implantitis in China. The main questions it aims to answer are:

* What is the prevalence of peri-implantitis in China
* What are the risk indicators of peri-implantitis in China

Participants will be invited to a free-of-charge clinical and radiographic examination of conventional dental implants present for over 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having at least one rough surface titanium implant in function for more than 5 years
2. Patients treated between January 1, 2013 and December 31, 2017
3. All the implants osseointegrated in the patients' mouth at the time of the examination (including those placed in external clinics) and having at least 5 years of loading, either proven by dental charts or confirmed by the patients, were evaluated

Exclusion Criteria:

1. Selected patients were invited to participate in the study by telephone calls on the numbers reported in their medical records, and if no response, the patient was not discarded until at least five attempts on different days have been made
2. Periapical and/or panoramic radiographs unavailable
3. History of peri-implantitis and/or peri-implant mucositis treatment
4. Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have conventional dental implants placed and over 5 years of functional loading.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-31 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Bleeding on probing [positive (+) or negative (-)] | About 5-10 years after surgery
  When bleeding is present after probing using a periodontal probe with a force of 0.2-0.3 N.
Peri-implant probing depth (mm) | About 5-10 years after surgery
  Measured using a periodontal probe inserted into the peri-implant sulcus
Bone loss (mm) | About 5-10 years after surgery
  Measured apically from the most coronal portion of the intraosseous part of the implant using periapical radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Yiqun Wu, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University